CLINICAL TRIAL: NCT01757977
Title: A Comparison of the Performance of Standard Double Lumen Tubes With Vivasight DL™ Double Lumen Tubes for Lung Isolation in Patients Undergoing Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Laffey (Other)
Responsible Party: Sponsor-Investigator, John Laffey, Professor of Anaesthesia and Critical Care, Consultant Anaesthetist, University College Hospital Galway
Organization: University College Hospital Galway (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C.A.751
Record Dates: First submitted 2012-12-22; First posted 2012-12-31 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Performance and Safety of an Airway Management Device
Keywords: Vivasight DL; double lumen endotracheal tube; fiberoptic confirmation of tube position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vivasight DL (Experimental): placement and intraoperative use of Vivasight DL double lumen endobronchial tube
  Interventions: Device: double lumen endotracheal tube placement and use
- standard DLT (Active Comparator): placement and intraoperative use of a standard double lumen endotracheal tube.
  Interventions: Device: double lumen endotracheal tube placement and use

INTERVENTIONS:
Device: double lumen endotracheal tube placement and use

SUMMARY:
The investigators have performed a number of studies on novel airway devices. In this randomized controlled trial he investigators would like to compare the performance of a new double-lumen endotracheal tube incorporating internal camera (Vivasight DL) with a standard double lumen tube.

DETAILED DESCRIPTION:
Single lung ventilation is frequently carried out to facilitate surgery on the lungs and pleura. In most instances this is achieved by insertion of a double-lumen endotracheal tube and then selectively ventilating one lung or both. Precise positioning of these tubes is essential for optimal performance. It has become the standard of care to perform bronchoscopy to confirm tube position.

A new double lumen endotracheal tube (Vivasight DL) has recently been developed. It has all the features of a standard double lumen endotracheal tube but also incorporates an internal camera which, when connected to an external screen, allows continuous confirmation of tube position.

This is randomized, single blinded controlled trial. The participants will be allocated to two study groups (Vivasight DL or standard DLT), in which the primary airway management device will be respectively Vivasight DL double lumen tube or a standard double lumen endotracheal tube.

Clinical Research Ethics Committee approval has been obtained. Suitable participants will be recruited after written informed consent.

Standard anesthetic preassessment and anesthesia will be provided.

Consenting patients passing the inclusion and exclusion criteria will be randomly allocated to either of the 2 study groups.

Protocol for attempts at placement and tube position confirmation will be followed.

The investigators will monitor a number of parameters, including time and ease of tube insertion, ability to verify tube position with the primary imaging modality for each group, need to perform tube position adjustment maneuvers, need to use fiberoptic bronchoscope during the case, quality of lung collapse, problems with ventilation and other.

The primary hypothesis is that the new Vivasight DL tube system will provide a comparable optical view to the fiberoptic scope view obtained via standard double lumen endotracheal tube in order to confirm optimal position.

ELIGIBILITY:
Inclusion Criteria:

* 16 - 85 yr old patients capable of informed consent
* ASA (American Society of Anesthesiologists physical status) 1-3
* non-emergency surgery of expected duration < 6 hours
* one-lung ventilation required

Exclusion Criteria:

* BMI > 35
* expected difficult airway
* Mallampati score >2
* increased risk of aspiration
* upper airway or upper GI problems
* live pregnancy

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Adequacy of optical view obtained to confirm optimal tube position. | within 60 minutes of commencement of general anesthesia
  The hypothesis is that the new Vivasight DL tube system will provide a comparable optical view to the fiberoptic scope view obtained via standard double lumen endotracheal tube in order to confirm optimal position.

SECONDARY OUTCOMES:
Time to confirmation of tube position | within 60 minutes of commencement of general anesthesia
Operator rated Device Difficulty Score | within 60 minutes of commencement of general anesthesia
  The investigators will use 10cm visual analogue scale (VAS) to rate the overall ease of device use till successful placement achieved and position confirmed optically.
Time from initial laryngoscopy to passing tube through vocal cords | Within 60 minutes of commencement of general anesthesia
rate of malposition | within 15 hours of commencement of general anesthesia
  the investigators will record the number/type of tube position adjustment maneuvers
need to pass a fiberoptic bronchoscope during case | within 15 hours of commencement of general anesthesia
presence of blood at the carina immediately post intubation | within 60 minutes of commencement of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Brian Harte, FFARCSI, Principal Investigator — Galway University Hospitals
Locations (1):
- Galway University Hospitals, Galway, Ireland